CLINICAL TRIAL: NCT03178929
Title: A Randomized Controlled Study on the Effect of S-Adenosyl Methionine Treatment on Anti-tumor Recurrence After Radical Treatment of Primary Hepatic Carcinoma
Brief Title: Effect of SAMe Treatment on Recurrence After Radical Treatment of Primary Hepatic Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Insight Science & Technology Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INW161116SAMe
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-Adenosyl Methionine Treatment (Experimental): Patients will be treated with S-Adenosyl Methionine treatment after radical treatment.
  2000mg, po
  Interventions: Drug: S-Adenosyl Methionine
- control group (No Intervention): Patients will be treated without S-Adenosyl Methionine treatment after radical treatment.

INTERVENTIONS:
Drug: S-Adenosyl Methionine — 2000mg, po
  Other Names: SAMe
  Arms: S-Adenosyl Methionine Treatment

SUMMARY:
The aim of this study is to explore the effect of SAMe on recurrence after radical treatment of Primary liver cancer.

DETAILED DESCRIPTION:
Primary liver cancer is now a major health problem. In the worldwide, PLC is the fifth most common cancer in male, the seventh in female, and has the second highest rate to cause death for men . Although the recent advances in treatment of Primary liver cancer have significantly improved the prognosis of patients with Primary liver cancer, the overall survival rate is still unsatisfactory. One of the reasons for the poor prognosis of Primary liver cancer is its high rate of recurrence. Anti-relapse treatment remains a pressing work to do.

In recent years, some study reported that SAMe had an impact on promoting apoptosis and inhibiting the growth on breast cancer, colon cancer, gastric cancer and liver cancer in vitro and vivo.

In this study, we aim to examine whether SAMe have an effect on improving patients' recurrence after radical treatment of Primary liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must sign the informed consent prior to the beginning of any study-related procedures;
* Patients diagnosed of Primary liver cancer;
* BCLC Stage：Stage 0、Stage A;
* Accept radical treatment;

Exclusion Criteria:

* With any other anti-cancer treatment before or after the surgery;
* Patients with extrahepatic metastasis;
* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction;
* Subjects accepting other trial drugs or participating in other clinical trials;
* Female with pregnancy or during the lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to tumor recurrence | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years

IPD SHARING:
Plan to Share IPD: Undecided